CLINICAL TRIAL: NCT07150936
Title: Effect of Stress Ball Intervention on Psychophysiological Responses During Hernia Surgery: A Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Muaz Gulsen, dr lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-SBF-CB-06
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hernia Surgery
Keywords: hernia surgery; stress ball; pain; Psychophysiological Response
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: There are 2 groups: control and intervention group
Who Masked: Participant, Outcomes Assessor
Masking Description: The intervention group will receive stress ball application during hernia surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants' demographic information will be collected interview using the Patient Information Form. Approximately 30 minutes before surgery, patients' systolic and diastolic blood pressure, heart rate, respiratory rate, and oxygen saturation will be measured and recorded. Pain severity will also be assessed using the VAS, and anxiety levels will be assessed using the VAS-A and Spielberger Trait Anxiety Scale.
  Intraoperative Period: All patients will be placed in the supine position on the operating room table. Patients in the intervention group will continue to use the stress ball for 15 minutes during the surgery, as per randomization. All patients will undergo a repeat 15-minute postoperative assessment of vital signs (systolic and diastolic blood pressure, heart rate, respiratory rate, oxygen saturation), pain with a VAS, and anxiety levels with a VAS-A.
  After the patients are taken to the clinic after the surgery, the same physiological measurements will repeated 10 mnt later
  Interventions: Behavioral: stress ball application
- no intervention group (No Intervention): Patients in the control group will only be treated with the clinic's current standard care protocol. Individuals in this group will not receive any additional interventions or stress ball applications. Measurements will be taken at the same timeframes and using the same methods as patients in the intervention group.

INTERVENTIONS:
Behavioral: stress ball application — Participants' demographic information will be collected interview using the Patient Information Form. Approximately 30 minutes before surgery, patients' systolic and diastolic blood pressure, heart rate, respiratory rate, and oxygen saturation will be measured and recorded. Pain severity will also be assessed using the VAS, and anxiety levels will be assessed using the VAS-A and Spielberger Trait Anxiety Scale. Intraoperative Period: All patients will be placed in the supine position on the operating room table. Patients in the intervention group will continue to use the stress ball for 15 minutes during the surgery, as per randomization. All patients will undergo a repeat 15-minute postoperative assessment of vital signs (systolic and diastolic blood pressure, heart rate, respiratory rate, oxygen saturation), pain with a VAS, and anxiety levels with a VAS-A. After the patients are taken to the clinic after the surgery, the same physiological measurements will repeated 10 mnt later
  Arms: intervention group

SUMMARY:
The aim of this study is to evaluate the effect of the stress ball applied during hernia surgery on the anxiety level, pain severity and vital signs of patients.

DETAILED DESCRIPTION:
Hernia surgery is a common procedure aimed at repairing hernias that develop in the abdominal and groin walls. Postoperative pain in repairs performed with synthetic mesh poses a significant problem, depending on surgical technique and individual factors. Preoperative pain level, psychological sensitivity, and previous surgical experience can influence the severity and duration of pain. Preoperative anxiety can trigger physiological and neuroendocrine responses, leading to intraoperative and postoperative complications, increased analgesic requirements, and decreased patient satisfaction. Nonpharmacological methods are recommended in addition to pharmacological treatments for acute pain management.These approaches not only reduce anxiety but also strengthen patient collaboration. One such method, the use of a stress ball, reduces pain and anxiety, increasing patient comfort. The literature indicates that stress balls reduce anxiety and stress levels, increase patient satisfaction, and positively impact vital signs. However, randomized controlled trials examining these effects in hernia surgery are limited. This research is expected to offer unique contributions to the applicability of nonpharmacological approaches in surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older,
* Willing to undergo surgery for an umbilical hernia, inguinal hernia, or femoral hernia,
* Have no hearing or perception problems,
* Have no physical disability that would prevent the use of a stress ball,
* Be undergoing hernia surgery for the first time.

Exclusion Criteria:

* Having used analgesic or anxiolytic medication before surgery,
* Being switched to general anesthesia during surgery despite planning for local anesthesia,
* Having a diagnosed psychiatric disorder,
* Being diagnosed with uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Spielberger State-Trait Anxiety Inventory | 5 months
  Developed by Spielberger and colleagues in 1970, this scale consists of two 20-item sections: the State Anxiety Inventory (STAI-I) and the Trait Anxiety Inventory (STAI-II). When assessing state anxiety, participants are asked to select one of the following options: "not at all," "a little," "a lot," or "completely." On the trait anxiety scale, responses are given as "almost never," "sometimes," "most of the time," or "most of the time." The scale's score ranges from 20 to 80, with higher scores indicating higher anxiety levels. In this study, the STAI-II scale will be administered preoperatively to assess patients' general anxiety levels and to identify differences in trait anxiety between groups.
Visual Anxiety Scale (VAS-A) | 5 months
  The Visual Anxiety Scale (VAS-A) is a simple, single-question measurement tool developed to assess individuals' anxiety levels. This method, long used in psychological analyses, is now widely used to assess pain, quality of life, and mood. The scale features a 10-centimeter horizontal line labeled "No anxiety" and "Very high anxiety." Patients mark the point on this line corresponding to their perceived anxiety level, and the distance between these marks is measured in millimeters to score the point. A higher measurement indicates a higher anxiety level. Despite its short length, the VAS-A is a tool with proven validity and reliability.
Visual Pain Scale (VAS) | 5 months
  Visual Pain Scale (VAS): The Visual Pain Scale (VAS) is a 10-cm-long line that can be applied horizontally or vertically to measure the level of pain experienced by an individual. The left end of the line is designated as "no pain," and the right end as "unbearable pain." The location of the point marked by the patient numerically reflects the intensity of the pain; the higher the score, the greater the perceived pain.
Vital Signs Monitoring Form | 5 months
  Vital Signs Monitoring Form: The Vital Signs Monitoring Form was developed based on a literature review to monitor the physiological parameters of patients undergoing hernia surgery. The form regularly records heart rate, systolic and diastolic blood pressure, respiratory rate, and oxygen saturation before, during, and after surgery. This allows for objective assessment of patients' hemodynamic status. Additionally, a Visual Pain Scale is included to measure pain levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Afsin State Hospital, Kahramanmaraş, Afşin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No